CLINICAL TRIAL: NCT03456583
Title: A Prospective Study To Evaluate The Performance And Operation Of The Brevera™ Breast Biopsy System
Brief Title: Brevera™ Breast Biopsy System Data Collection Study
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-05A
Record Dates: First submitted 2018-02-20; First posted 2018-03-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Female
Keywords: Breast Biopsy; Breast Biopsy Imaging; Stereotactic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Brevera Breast Biopsy System: The Brevera Breast Biopsy System with CorLumina imaging technology is a vacuum-assisted biopsy device, which is used to remove breast tissue in a minimally invasive manner using stereotactic or tomosynthesis imaging. A breast biopsy is a test that removes tissue or sometimes fluid from the suspicious area. The removed cells are examined under a microscope and further tested to check for the presence of breast cancer. A biopsy is a diagnostic procedure that can definitely determine if the suspicious area is cancerous.
  Interventions: Device: Brevera Breast Biopsy System

INTERVENTIONS:
Device: Brevera Breast Biopsy System — The Brevera Breast Biopsy System with CorLumina imaging technology is a vacuum-assisted biopsy device, which is used to remove breast tissue in a minimally invasive manner using stereotactic or tomosynthesis imaging. A breast biopsy is a test that removes tissue or sometimes fluid from the suspicious area. The removed cells are examined under a microscope and further tested to check for the presence of breast cancer. A biopsy is a diagnostic procedure that can definitely determine if the suspicious area is cancerous.

SUMMARY:
The Brevera Breast Biopsy System integrates tissue acquisition, real time imaging, and post biopsy handling all during the same procedure. This post-market clinical trial will be performed to obtain clinical/operational data and feedback on the Brevera Breast Biopsy System.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years of age or older
* Subject has at least one breast imaging finding requiring biopsy for which images are available
* Subject is able to understand, read and sign the trial specific informed consent form after the nature of the trial has been fully explained to her

Exclusion Criteria:

* Patients who, based on the physician's judgment, may be at increased risk or develop complications associated with core removal or biopsy.
* Patients receiving anticoagulant therapy or may have bleeding disorders which may put the patient at increased risk of procedural complications based upon physicians judgment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any woman who is scheduled for a stereotactic breast biopsy (for possible breast cancer) who meets the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Keller, Study Director — Hologic, Inc.
Locations (6):
- Institut régional du Cancer de Montpellier, Montpellier, France
- Brustdiagnostik Munchen, Tübingen, Germany
- Radiologia Senologica, Milan, Italy
- Noordwest Ziekenhuisgroep, Alkmaar, Netherlands
- Centro de Patalogia de la Mama-Fundacion Tejerina, Madrid, Spain
- Royal Free Londan NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brevera Breast Biopsy System
Started | 500
Completed | 500
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brevera Breast Biopsy System
Number analyzed (Participants) | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 500
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 57.4 [33 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 500
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 100
  United Kingdom | 91
  Italy | 100
  France | 81
  Germany | 28
  Spain | 100

OUTCOME MEASURES:

1. Primary Outcome: Procedural Time
Description: Total time elapsed between from when the subject enters the procedure room until she has left the procedure room.
Time Frame: Through study completion, enrollment expected to take up to 6-10 months at each site - Data collected from day of Breast Biopsy Procedure Only
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Brevera Breast Biopsy System
Number analyzed (Participants) | 500
Minutes | 38.44 (14.17)

2. Secondary Outcome: Post-biopsy Complication Rates
Description: Adverse event rates.
Time Frame: as for outcome 1
Population: Enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Brevera Breast Biopsy System
Number analyzed (Participants) | 500
Participants | 11

3. Secondary Outcome: Average Number of Cores Per Lesion
Description: The average number of cores obtained for each lesion across all sites.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: Cores Per Lesion
Units Other Than Participants: lesions
Arm/Group | Brevera Breast Biopsy System
Number analyzed (Participants) | 500
Number analyzed (lesions) | 530
Cores Per Lesion | 10.58 [2 to 48]

4. Secondary Outcome: Percentage of Procedures With Overall Positive Opinion From Radiologist, Technologist, and Patient
Description: The radiologists, technologists, and patients participating in this study were asked to provide feedback on the Brevera Biopsy System at the completion of each procedure. Their responses (raw scores) were reported and converted to percentage of procedures with overall positive opinions. The scale goes from 0% (poor/negative opinion) to 100% (excellent/positive opinion).
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: Percentage of procedures
Groups:
- Radiologists' Feedback: Radiologist positive overall opinion of the Brevera Biopsy System for the procedures (scored 1-5 on Likert Scale).
- Technologists' Feedback: Technologist with a positive overall opinion of the Brevera Biopsy System for the proceudres (scored 1-5 on Likert Scale).
- Patients' Feedback: Patient agreed that they were satisfied with the facility and the care that they received during the procedure (scored 1-5 on Likert Scale).
Arm/Group | Radiologists' Feedback | Technologists' Feedback | Patients' Feedback
Number analyzed (Participants) | 497 | 496 | 496
Percentage of procedures | 76.3 [8.45 to 91.5] | 66.9 [10.1 to 89.9] | 96.8 [0.6 to 99.4]

ADVERSE EVENTS:
Time Frame: subjects were evaluated for the time the procedure began to the release from the outpatient treatment facility per standard of care for any adverse events that they experienced.
Description: There was no Serious Adverse Event There was no Mortality
Arm/Group | Brevera Breast Biopsy System
All-Cause Mortality (participants affected / at risk) | 0/500
Serious Adverse Events (participants affected / at risk) | 0/500
Other Adverse Events (participants affected / at risk) | 11/500
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brevera Breast Biopsy System (N=500)
Hematoma (Injury, poisoning and procedural complications) | 9
Excessive Bleeding (Injury, poisoning and procedural complications) | 1
Dislocation of the marker due to some of the postprocedure haemorrage (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT03456583/Prot_SAP_000.pdf